CLINICAL TRIAL: NCT03251612
Title: Predictive Value of In-vitro Testing Anti-cancer Therapy Sensitivity on Tumorspheres From Patients With Metastatic Colorectal Cancer
Brief Title: Predictive Value of Drug Sensitivity Testing Tumorspheres From Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tumorspheres Colrec
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Other): 1 drug or a combination of drugs considered standard anticancer treatment is given according to the result of the sensitivity analysis.
  Interventions: Drug: Based on sensitivity analysis

INTERVENTIONS:
Drug: Based on sensitivity analysis — * 5FU, infusional
  * Capecitabine
  * Oxaliplatin (FOLFOX)
  * Irinotecan (FOLFIRI)
  * FOLFOXIRI (triplet)
  * Bevacizumab
  * Panitumumab
  * Cetuximab
  * Regorafenib
  * Tas-102
  * Ramucirumab
  * Aflibercept
  * Pembrolizumab
  * Nivolumab
  * Vinorelbine and capecitabine
  * Sorafenib
  * Gemcitabine and capecitabine
  * Olaparib
  * Epirubicin

SUMMARY:
The purpose of the present study is to investigate the benefit of anti-cancer therapy administered on the basis of drug sensitivity testing. This concerns colorectal cancer patients who have previously received standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer

  * Biopsy proven adenocarcinoma compatible with colorectal origin (primary tumor or metastasis)
  * If only biopsy from metastasis can be obtained, the patient must have a previously resected or image proven tumor of the colon or rectum (scanning or endoscopy)
  * Non-resectable metastatic spread
* Previously exposed to or intolerance or contraindications to standard systemic therapy, defined as

  * oxaliplatin
  * irinotecan
  * 5-fluorouracil (or similar such as capecitabine, S1)
  * VEGF inhibitor bevacizumab
  * EGFR inhibitor panitumumab or cetuximab (if RAS/RAF wt)
* Progressive disease defined as progression according to RECIST 1.1
* ECOG performance status 0-2
* Age at least 18 years
* Adequate bone marrow, liver and renal function allowing systemic chemotherapy

  * Absolute neutrophil count ≥1.5x10^9/l and thrombocytes ≥ 100x10^9/l.
  * Bilirubin ≤ 1.5 x upper normal value and alanine aminotransferase ≤ 3 x upper normal value
  * Calculated or measured renal glomerular filtration rate at least 30 mL/min
* Anticonception for fertile women and for male patients with a fertile partner. Intrauterine device, vasectomy of a female subject's male partner or hormonal contraceptive are acceptable
* Written and orally informed consent

Exclusion Criteria:

* Incapacity, frailty, disability, or comorbidity to a degree that according to the investigator is not compatible with participation in the protocol
* Other active malignant disease requiring therapy
* Other systemic anti-cancer therapy (palliative radiotherapy is allowed).
* Pregnant (positive pregnancy test) or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2021-08-23 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Progression free survival 8 weeks after start of treatment | 42-63 days after start of treatment

SECONDARY OUTCOMES:
Progression free survival | Every 8 weeks until progression or death up to 2.5 years
Overall survival | Every 3 months up to 2.5 years
Response rate | Every 8 weeks until progression up to 2.5 years
Quality of life as measured by questionnaire EQ-5D-5L | Every 8 weeks up to 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars H Jensen, MD, Study Chair — Vejle Hospital
Locations (4):
- Denmark (3):
  - Department of Oncology, Aalborg University Hospital, Aalborg
  - Department of Oncology, Rigshospitalet, Copenhagen
  - Departmen of Oncology, Vejle Hospital, Vejle
- Universitätsklinikum Hamburg - Eppendorf, Universitäres Cancer Center Hamburg (UCCH), Hamburg, Germany

REFERENCES:
- [Derived] Jensen LH, Rogatto SR, Lindebjerg J, Havelund B, Abildgaard C, do Canto LM, Vagn-Hansen C, Dam C, Rafaelsen S, Hansen TF. Precision medicine applied to metastatic colorectal cancer using tumor-derived organoids and in-vitro sensitivity testing: a phase 2, single-center, open-label, and non-comparative study. J Exp Clin Cancer Res. 2023 May 5;42(1):115. doi: 10.1186/s13046-023-02683-4. PMID 37143108